CLINICAL TRIAL: NCT03861299
Title: The SAFE-Trial: Safe Surgery for Glioblastoma Multiforme: Awake Craniotomy Versus Surgery Under General Anesthesia. A Multicenter Prospective Randomised Controlled Study
Brief Title: The SAFE-Trial: Awake Craniotomy Versus Surgery Under General Anesthesia for Glioblastoma Patients.
Acronym: SAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jasper Gerritsen (Other)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other); University Medical Center Groningen (Other); Medical Center Haaglanden (Other); University Hospital, Ghent (Other)
Responsible Party: Sponsor-Investigator, Jasper Gerritsen, Study Coordinator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL66673.078.18; MEC-2018-1564 (Other: Medical Ethical Committee Erasmus MC)
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioblastoma Multiforme of Brain; Astrocytoma, Grade IV; Brain Tumor; Brain Cancer; Brain Neoplasms
Keywords: Glioblastoma; Neurological morbidity; Postoperative complications; Extent of resection; Gross-total resection; Health-related quality of life; Progression-free survival; Overall survival
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Each participating center will randomise eligible and willing patients through the webbased clinical database and randomisation application ALEA. The Clinical Trial Centre (CTC) of the Erasmus MC will build the randomisation application by use of a dynamic allocation algorithm (minimization), in which patients are allocated to keep the imbalance between treatment groups to a minimum at every stage of recruitment within the covariates age (≤55 years vs >55years), Karnofsky performance scale (80-90 vs >90), and left or right hemisphere. Treatment allocation and allocated subject number will be shown immediately on screen and will in addition automatically be emailed to local investigators and other study personnel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awake craniotomy (Experimental): Cortical stimulation is performed with a bipolar electrical stimulator. The Boston naming test and repetition of words is done in cooperation with a neuropsychologist/linguist, who will inform the neurosurgeon of any kind of speech arrest or dysarthria. When localizing the motor and sensory cortex, the patient is asked to report any unintended movement or sensation in extremities or face. Functional cortical areas are marked with a number. When the tumour margins or white matter is encountered or when on regular neuronavigation the eloquent white matter tracts are thought to be in close proximity, subcortical stimulation (biphasic currents of 8-16 mA, pulse frequency 60 Hz, single pulse phase duration of 100 microsec., 2-second train) is performed to localize functional tracts.
  Interventions: Procedure: Awake craniotomy
- Craniotomy under general anesthesia (Active Comparator): Trephination and tumour resection are performed without any additional neuro-psychological monitoring or brain mapping, guided by STEALTH-neuronavigation.
  Interventions: Procedure: Craniotomy under general anesthesia

INTERVENTIONS:
Procedure: Awake craniotomy — Awake craniotomy
  Other Names: Intraoperative stimulation monitoring with (sub)cortical electrostimulation; Intraoperative brain mapping with (sub)cortical electrostimulation
  Arms: Awake craniotomy
Procedure: Craniotomy under general anesthesia — Craniotomy under general anesthesia
  Arms: Craniotomy under general anesthesia

SUMMARY:
The trial is designed as a multicenter randomized controlled study. 246 patients with presumed Glioblastoma Multiforme in eloquent areas on diagnostic MRI will be selected by the neurosurgeons according the eligibility criteria (see under). After written informed consent is obtained, the patient will be randomized for an awake craniotomy (AC) (+/-123 patients) or craniotomy under general anesthesia (GA) (+/-123 patients), with 1:1 allocation ratio. Under GA the amount of resection of the tumour has to be performed within safe margins as judged by the surgeon during surgery. The second group will be operated with an awake craniotomy procedure where the resection boundaries for motor or language functions will be identified by direct cortical and subcortical stimulation. After surgery, the diagnosis of GBM will have to be histologically confirmed. If GBM is not histologically confirmed, patients will be considered off-study and withdrawn from the study. These patients will be followed-up according to standard practice. Thereafter, patients will receive the standard treatment with concomitant Temozolomide and radiation therapy and standard follow up. Total duration of the study is 5 years. Patient inclusion is expected to take 4 years. Follow-up is 1 year after surgery. Statistical analysis, cost benefit analysis and article writing will take 3 months.

DETAILED DESCRIPTION:
Rationale Glioblastoma Multiforme (GBM) or Astrocytoma's grade IV (WHO) are devastating tumors with one of the worst prognoses in oncology. Extending resection improves survival in patients with GBM. Surgery of GBM nowadays is usually performed under general anesthesia (GA) and resections are not as aggressive as possible, due to the chance of seriously damaging the patient with a rather low life expectancy. A surgical technique optimizing resection of the tumor in eloquent areas but preventing neurological deficits is necessary to improve survival and quality of life in these patients. Awake craniotomy (AC) with the use of cortical and subcortical stimulation is an alternative surgical technique that is standardly implemented in surgery for low grade glioma, but not yet for GBM. AC has shown to increase resection percentage and preserve quality of life in low grade glioma (LGG) and could be of important value in the surgery of GBM.

Objective The study is performed to increase safety and efficacy during surgery in patients with GBM in eloquent areas. This study will compare awake craniotomy with surgery under general anesthesia for patients with GBM near or in eloquent areas. Primary end points are: 1) Proportion of patients with NIH Stroke Scale (NIHSS) deterioration at 6 weeks post- surgery, where deterioration is defined as at least one point increase in total NIHSS score compared to baseline. 2) Proportion of patients without residual contrast-enhancing tumour on postoperative MRI. Secondary end points are: 1) Health related quality of life (HRQoL) at 6 weeks, 3 months and 6 months after operation. 2) Progression-free survival (PFS) at 12 months after operation. 3) Overall survival (OS) at 12 months after operation. 4) Frequency and severity of Serious Adverse Effects in each group: Infections, intracranial bleeding, epilepsy, aphasia, paresis/paralysis in arms or/and legs. Also, a cost benefit analysis will be performed.

Study design The trial is set up as a multicenter randomized controlled study. The study will include 246 patients in 5 neurosurgical centers in the Netherlands. Patients with GBM in eloquent areas on diagnostic MRI will be selected by the neurosurgeons according to the eligibility criteria. After informed consent the patient will be randomized for awake craniotomy (AC) or regular craniotomy under general anesthesia (GA) with 1:1 allocation ratio. After surgery, only patients with histologically proven GBM will continue with the study. Patients in whom no GBM could not be proven histologically, will be considered off-study. Thereafter, patients will receive the standard treatment with concomitant Temozolomide and radiation therapy and standard follow up. Total duration of the study is 5 years. Patient inclusion is 4 years. Follow-up is 1 year.

Study population Patients aged 18-90 years old, with Glioblastoma Multiforme near or in eloquent areas and eligible for awake craniotomy.

Intervention Awake craniotomy compared to craniotomy under general anaesthesia

Main study parameters/endpoints

1. Proportion of patients with NIHSS deterioration at 6 weeks post-surgery
2. Proportion of patients without residual contrast-enhancing tumour on postoperative MRI

Nature and extent of the burden and risks associated with participation, benefit and group relatedness Patients have 50% chance to be randomized for an awake procedure. The risk-benefit-ratio of this procedure in patients with GBM is subject of this trial and the investigators expect less neurological morbidity than surgery under generalised anaesthesia. Three quality of life questionnaires and 1 neurological examination will take place preoperatively, 6 weeks after, 3 months after and 6 months after the surgery. The burden of this trial for the patient is therefore confined.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 90 years
2. Tumor diagnosed as Glioblastoma Multiforme on MRI with distinct ring-like pattern of contrast enhancement with thick irregular walls and a core area reduced signal suggestive of tumour necrosis as assessed by the surgeon
3. Tumors situated in or near eloquent areas; motor cortex, sensory cortex, subcortical pyramidal tract or speech areas as indicated on MRI (Sawaya Grading II and II)
4. The tumor is suitable for resection (according to neurosurgeon)
5. Karnofsky performance scale 80 or more
6. Written Informed consent

Exclusion Criteria:

1. Tumors of the cerebellum, brain stem or midline
2. Multifocal contrast enhancing lesions
3. Substantial non-contrast enhancing tumor areas suggesting low grade gliomas with malignant transformation
4. Medical reasons precluding MRI (eg, pacemaker)
5. Inability to give consent because of or language barrier
6. Psychiatric history
7. Previous brain tumour surgery
8. Previous low-grade glioma.
9. Second primary malignancy within the past 5 years with the exception of adequately treated in situ carcinoma of any organ or basal cell carcinoma of the skin.
10. Severe aphasia or dysphasia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative neurological morbidity | Between operation and 6 weeks postoperatively
  Proportion of patients with NIHSS (National Institute of Health Stroke Scale) deterioration at 6 weeks post-surgery, where deterioration is defined as at least one point increase in total NIHSS score compared to baseline
Proportion of gross-total resections | Assessed on 48 hours postoperative scan
  Proportion of patients without residual contrast-enhancing tumour on postoperative MRI, where residual tumour is defined as contrast-enhancement with a volume more than 0.175 cm3.

SECONDARY OUTCOMES:
Health-related quality of life assessed by EQ-5D questionnaire | Between baseline and 6 weeks/3 months/6 months postoperatively
  Health related quality of life (HRQoL) at 6 weeks, 3 and 6 months after operation, where HRQol is measured with the EQ-5D questionnaire
Health-related quality of life assessed by EORTC-QLQ-BN20 questionnaire | Between baseline and 6 weeks/3 months/6 months postoperatively
  Health related quality of life (HRQoL) at 6 weeks, 3 and 6 months after operation, where HRQol is measured with the EORTC QLQ-BN20 questionnaire
Health-related quality of life assessed by EORTC-QLQ-C30 questionnaire | Between baseline and 6 weeks/3 months/6 months postoperatively
  Health related quality of life (HRQoL) at 6 weeks, 3 and 6 months after operation, where HRQol is measured with the EORTC-QLQ-C30 questionnaire
Progression-free survival | Between surgery and 12 months postoperatively
  Progression-free survival (PFS) at 12 months defined as time from diagnosis to disease progression (occurrence of a new tumour lesion with a volume greater than 0.175 cm3, or an increase in residual tumour volume of more than 25%) or death, whichever comes first
Overall survival | Between surgery and 12 months postoperatively
  Overall survival (OS) at 12 months defined as time from diagnosis to death from any cause
Postoperative (serious) adverse events | Between surgery and 6 weeks postoperatively
  Frequency and severity of (Serious) Adverse Effects in each group: Infections, intracerebral hemorrhage, epilepsy, aphasia, paresis/paralysis in arms or/and legs

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Vincent, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- University Hospital Ghent, Ghent, Belgium
- Netherlands (4):
  - Elisabeth-Tweesteden Ziekenhuis, Tilburg, North Brabant
  - Erasmus MC, Rotterdam, South Holland
  - Medical Center Haaglanden, The Hague, South Holland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gerritsen JKW, Zwarthoed RH, Kilgallon JL, Nawabi NL, Jessurun CAC, Versyck G, Pruijn KP, Fisher FL, Lariviere E, Solie L, Mekary RA, Satoer DD, Schouten JW, Bos EM, Kloet A, Nandoe Tewarie R, Smith TR, Dirven CMF, De Vleeschouwer S, Broekman MLD, Vincent AJPE. Effect of awake craniotomy in glioblastoma in eloquent areas (GLIOMAP): a propensity score-matched analysis of an international, multicentre, cohort study. Lancet Oncol. 2022 Jun;23(6):802-817. doi: 10.1016/S1470-2045(22)00213-3. Epub 2022 May 12. PMID 35569489
- [Derived] Gerritsen JKW, Dirven CMF, De Vleeschouwer S, Schucht P, Jungk C, Krieg SM, Nahed BV, Berger MS, Broekman MLD, Vincent AJPE. The PROGRAM study: awake mapping versus asleep mapping versus no mapping for high-grade glioma resections: study protocol for an international multicenter prospective three-arm cohort study. BMJ Open. 2021 Jul 21;11(7):e047306. doi: 10.1136/bmjopen-2020-047306. PMID 34290067
- [Derived] Gerritsen JKW, Klimek M, Dirven CMF, Hoop EO, Wagemakers M, Rutten GJM, Kloet A, Hallaert GG, Vincent AJPE. The SAFE-trial: Safe surgery for glioblastoma multiforme: Awake craniotomy versus surgery under general anesthesia. Study protocol for a multicenter prospective randomized controlled trial. Contemp Clin Trials. 2020 Jan;88:105876. doi: 10.1016/j.cct.2019.105876. Epub 2019 Oct 30. PMID 31676314